CLINICAL TRIAL: NCT02992964
Title: Pilot Study of Nivolumab in Pediatric Patients With Hypermutant Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawal of drug supply/funding
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Daniel Morgenstern, Staff Oncologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-075
Record Dates: First submitted 2016-12-02; First posted 2016-12-14 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Refractory or Recurrent Hypermutated Malignancies; Biallelic Mismatch Repair Deficiency (bMMRD) Positive Patients
MeSH Terms: conditions — Turcot syndrome | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Regimen: Nivolumab will be administered every 14 days until disease progression or treatment discontinuation due to unacceptable toxicities. Treatment may extend up to 2 years in patients who show clinical and radiological benefit.
  Dose: 3 mg/kg intravenously as a continuous infusion over 60 min (+/-10 min window)
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab (also referred to as BMS-936558 or MDX1106) is a human monoclonal antibody (HuMAb; immunoglobulin G4 [IgG4]-S228P) that targets the programmed death-1 (PD-1) cluster of differentiation 279 (CD279) cell surface membrane receptor.
  Other Names: OPDIVO

SUMMARY:
This is an open-label, single arm, multi-center, pilot study of Nivolumab in pediatric patients with recurrent or refractory hypermutant malignancies aged 12 months to 18 years of age. This study is to assess clinical and radiological benefits of treatment with Nivolumab in children with hypermutated cancers, including those with bMMRD syndrome. It is our expectation that patients with bMMRD syndrome will account for the majority of patients enrolled on this study.

ELIGIBILITY:
Inclusion Criteria:

Part I

1. Consent/ Assent: Patient and/or Legally Acceptable Representative (LAR; such as a parent or guardian, as applicable) must be willing and able to provide written informed consent/assent for the trial as per local requirements.
2. Age: patients must be ≥ 12 months and <25 years of age at time of Part I enrollment. Local centres are only obligated to treat/ admit patients in accordance their age range capabilities.
3. Recurrent or relapse paediatric cancer patients suspected to be hypermutant, including those exhibiting evidence of one or more of the following:

   1. high microsatellite instability (MSI-H) in current or previous tumour;
   2. a mutation causing loss of mismatch repair gene (MLH1, MSH2, MSH6, PMS2, EPCAM or MSH3) expression;
   3. hypermutation by local sequencing in current or previous tumour;
   4. a history of CMMRD, Lynch syndrome, xeroderma pigmentosum (XP), or other established disorder affiliated with an elevated hypermutation rate;
   5. a functional mutation of polymerase genes (POLE or POLD1) in current or previous tumour;
   6. a functionally impaired RRD pathway by other means;
   7. a temozolomide (TMZ) treated current or previous CNS tumour;
   8. a predisposing hypermutant cancer signature (i.e. dysregulation of an apolipoprotein B mRNA editing enzyme, catalytic polypeptide-like (APOBEC) cytidine deamination or UV-associated);
   9. other factors, which may predicate an elevated mutation burden at the discretion of the Study Chair or Co-Chair.
4. Diagnosis: patients must have histologic or cytologic confirmation of malignancy at the time of initial diagnosis or relapse (as specified above). Patients with multiple concurrent and/or sequential neoplasms are eligible, including CNS and haematological malignancies.
5. Specimen availability: patients must be able to provide specimen (archival or newly obtained biopsy) of a tumor lesion, appropriately obtained and preserved in a manner compatible for TMB analysis or applicable IHC staining for MMR gene protein expression, if applicable (as described in the Lab Manual). Only those with an already ascertained TMB level report from the laboratory specified in the Lab Manual or those with proof of RRD as outlined in the Lab Manual will be exempt from mandatory tissue submission.

If tissue (including archival) is not available, a new tissue specimen may be obtained if deemed clinically appropriate. Any such biopsy will not be considered a trial-related procedure.

Inclusion Criteria Part II

1. Consent/ Assent: Patient and Legally Acceptable Representative (LAR; such as a parent or guardian, as applicable) must be willing and able to provide written informed consent/assent for the trial as per local requirements.
2. Confirmation of hypermutation or Proof of RRD: patient must have completed and verified a sufficient TMB level or have proof of RRD diagnosed in the appropriate lab, as outlined in the Lab Manual.
3. Age: patients must be ≥ 12 months and < 25 years of age at the time of Part II enrollment. Local centres are only obligated to treat/ admit patients in accordance their age range capabilities.
4. Diagnosis: patients must have had histologic verification of malignancy at the time of initial diagnosis or at relapse (as specified above). Patients with multiple concurrent and/or sequential neoplasms are eligible, including CNS and haematological malignancies.
5. Disease status: patients must have either measurable or evaluable disease in accordance with criteria as outlined in Section 10. Tumour lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Treatment options: patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life. Chemotherapy-naïve patients will be eligible in cases where first-line therapy does not include chemotherapy (e.g. surgery alone for management of ependymoma).
7. Performance status: Karnofsky ≥ 50% for patients > 16 years of age or Lansky ≥ 50 for patients ≤ 16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
8. Previous treatment: patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy.

   1. Myelosuppressive chemotherapy: at least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea).
   2. Hematopoietic growth factors: at least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the Study Chair or Co-Chair.
   3. Biologic (anti-neoplastic agent): at least 14 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 14 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the Study Chair or Co-Chair.
   4. Monoclonal antibodies: at least three (3) half-lives of the antibody after the last dose of a monoclonal antibody.
   5. Radiation Therapy (XRT): at least 14 days after local palliative XRT (small port). At least 150 days must have elapsed if prior Total Body Irradiation, craniospinal XRT or if ≥ 50% radiation of pelvis. At least 42 days must have elapsed if other substantial BM radiation.
   6. Stem Cell Infusion without Total Body Irradiation (TBI): no evidence of active graft vs. host disease and at least 56 days must have elapsed after transplant or stem cell infusion. Patients with prior allogeneic transplants (including solid organ) are not eligible.
9. Organ Function Requirements:

   a. Adequate BM Function Defined as i. Peripheral absolute neutrophil count (ANC) ≥0.75 x 109/L or 750/mm3. ii. Platelet count ≥75 x 109/L or 75,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment.

   iii. Hemoglobin ≥ 90g/L (transfusion permitted). iv. Patients with known BM metastatic disease or haematological malignancies will be eligible for study provided they meet haematological criteria. These patients may receive transfusions (e.g. to achieve platelet threshold) provided they are not known to be refractory to platelet transfusions but will not be evaluable for hematologic toxicity.

   b. Adequate Renal Function Defined as: A serum creatinine based on age/gender as provided in Table 3 (see Section 4.2.2) c. Adequate Liver Function Defined as: i. Bilirubin (sum of conjugated + unconjugated or total bilirubin) ≤1.5x institutional upper limit of normal (ULN) for age (except for patients with Gilbert's Syndrome, when bilirubin of < 51 µmol/L or 3.0 mg/dL is permitted).

   ii. ALT/AST:

1. ≤ 2.5 x institutional ULN for patients without liver metastases. 2. ≤ 5 x institutional ULN for patients with liver metastases. d. Adequate Pulmonary Function Defined as: No history of chronic pulmonary disease (such as Cystic Fibrosis) and no evidence of dyspnea at rest, no exercise intolerance due to pulmonary insufficiency and a pulse oximetry > 92% on room air.

e. Adequate Pancreatic Function Defined as: Serum lipase ≤ ULN. Patients with glucose intolerance should be on a stable regiment and be monitored.

10. For patients with brain tumors, debulking surgery prior to treatment with nivolumab should be considered when appropriate to reduce the risk of pseudoprogression-associated toxicities. Such debulking surgery is not mandatory for trial enrollment. Patients should be recovered from surgery and wait at least 7 days from surgery before first dose.

Exclusion Criteria:

Part II Only

1. Women who are pregnant or breastfeeding and men who are sexually active with women of childbearing potential (WOCBP)* who are not willing to use effective contraception, or to practice abstinence if this is the usual lifestyle and preferred contraception for the patient. **

   * Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as there is yet no available information regarding human fetal or teratogenic toxicities.
   * WOCBP must have a negative serum pregnancy test every 4 weeks. and During Part II screening, WOCBP must have a negative serum pregnancy test. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab administration. WOCBP who are sexually active, must be willing to adhere to effective contraception during treatment and for 5 months after the last dose of nivolumab.
   * Men who are sexually active with WOCBP must be willing to adhere to effective contraception during treatment and for 7 months after the last dose of nivolumab.
   * Women who are surgically sterile, as well as azoospermic men do not require contraception.
2. Concomitant Medications

   1. Corticosteroids: Patients requiring systemic steroid therapy or any other form of immunosuppressive therapy within seven (7) days prior to first dose of trial therapy or while on trial are not eligible. The use of physiologic doses of corticosteroids (up to 5mg/m2/day prednisone equivalent) is permitted following discussion with the Study Chair or Co-Chair.
   2. Investigational Drugs: Patients who are currently receiving another investigational drug are not eligible.
   3. Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents are not eligible.
3. Patients with a History of Autoimmune Disease

   • Patients with a history of autoimmune disorder that has required systemic treatment in the previous two (2) years are not eligible. Asymptomatic laboratory abnormalities (e.g. ANA, rheumatoid factor, altered thyroid function studies) will not render a patient ineligible in the absence of a diagnosis of an autoimmune disorder. Replacement therapy (e.g. thyroxine, insulin or physiologic corticosteroid replacement therapy) is not considered a form of systemic treatment.
4. Infection: Patients who have an uncontrolled infection are not eligible.
5. HIV and/or Hepatitis B/C patients: Patients with known HIV/AIDS or acute/chronic Hepatitis B or C are excluded.
6. Transplant patients: Patients who have received prior allogeneic Bone Marrow (BM) transplants or prior solid organ transplantation are not eligible.
7. Non-Compliance: Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.
8. Previous anti-PD-1 and/or anti-PD-L1 therapy: Patients who have received prior anti-PD-1 and/or anti-PD-L1 directed therapy (mAb or small molecule) are not eligible.
9. Live vaccines: Patients who have received a live vaccine within 30 days of start of study treatment are not eligible.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
To evaluate the objective response rate to Nivolumab in bMMRD positive pediatric patients with refractory hypermutated malignancies | 5 years (60 months) from date of enrollment
  Objective response rate will assessed by physical assessments, lab values, disease assessments and adverse events that are related to treatment. Scheduled time-points and the above assessments are detailed further in section "9.1 Study Calendar" of the protocol.
To evaluate the objective response rate to Nivolumab in bMMRD positive pediatric patients with recurrent hypermutated malignancies. | 5 years (60 months) from date of enrollment
  Objective response rate will assessed by physical assessments, lab values, disease assessments and adverse events that are related to treatment. Scheduled time-points and the above assessments are detailed further in section "9.1 Study Calendar" of the protocol.
Estimating the feasibility of using Nivolumab as a treatment in bMMRD positive, pediatric patients with refractory or recurrent hypermutated malignancies. | 5 years (60 months) from date of enrollment
  Feasibility of treatment will be measured using a patient's disease response assessment. This means using standard RECIST criteria for solid tumours, iRANO/RANO criteria for CNS malignancies and the revised AML International Working Group (IWG) Criteria for haematological malignancies; modified RECIST criteria for immune response may be considered during the time of study.

SECONDARY OUTCOMES:
The progression free survival (PFS) of pediatric patients with progressive or recurrent hypermutated malignancies including bMMRD patients treated with Nivolumab. | 5 years (60 months) from date of enrollment
Number of Participants with Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 5 years (60 months) from date of enrollment
  These will be assessed by abnormal findings in physical assessments, lab values, disease assessments and adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Morgenstern, MB BChir PhD, Principal Investigator — The Hospital for Sick Children
Locations (10):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Australia (3):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
- Canada (2):
  - Children's & Women's Health Centre of British Columbia, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario
- France (2):
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif
- Tel Aviv Sourasky Medical Centre, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Das A, Tabori U, Sambira Nahum LC, Collins NB, Deyell R, Dvir R, Faure-Conter C, Hassall TE, Minturn JE, Edwards M, Brookes E, Bianchi V, Levine A, Stone SC, Sudhaman S, Sanchez Ramirez S, Ercan AB, Stengs L, Chung J, Negm L, Getz G, Maruvka YE, Ertl-Wagner B, Ohashi PS, Pugh T, Hawkins C, Bouffet E, Morgenstern DA. Efficacy of Nivolumab in Pediatric Cancers with High Mutation Burden and Mismatch Repair Deficiency. Clin Cancer Res. 2023 Dec 1;29(23):4770-4783. doi: 10.1158/1078-0432.CCR-23-0411. PMID 37126021
- [Derived] Henderson JJ, Das A, Morgenstern DA, Sudhaman S, Bianchi V, Chung J, Negm L, Edwards M, Kram DE, Osborn M, Hawkins C, Bouffet E, Cho YJ, Tabori U. Immune Checkpoint Inhibition as Single Therapy for Synchronous Cancers Exhibiting Hypermutation: An IRRDC Study. JCO Precis Oncol. 2022 Mar;6:e2100286. doi: 10.1200/PO.21.00286. No abstract available. PMID 35235414
- [Derived] Rittberg R, Harlos C, Rothenmund H, Das A, Tabori U, Sinha N, Singh H, Chodirker B, Kim CA. Immune Checkpoint Inhibition as Primary Adjuvant Therapy for an IDH1-Mutant Anaplastic Astrocytoma in a Patient with CMMRD: A Case Report-Usage of Immune Checkpoint Inhibition in CMMRD. Curr Oncol. 2021 Feb 1;28(1):757-766. doi: 10.3390/curroncol28010074. PMID 33535600